CLINICAL TRIAL: NCT00003315
Title: Supplementary Protocol for Patients With Invasive Fungal Infection, Entered Into AML 11, AML 12 and UKALL XII (Or Their Successors)
Brief Title: Liposomal Amphotericin B With or Without Sargramostim in Treating Patients With Invasive Fungal Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: CDR0000066264; MRC-LEUK-IFI; EU-97030
Record Dates: First submitted 1999-11-01; First posted 2004-08-26 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2007-05

CONDITIONS: Infection
Keywords: infection
MeSH Terms: conditions — Infections | interventions — sargramostim; liposomal amphotericin B

INTERVENTIONS:
Biological: sargramostim
Drug: liposomal amphotericin B

SUMMARY:
RATIONALE: Drugs like liposomal amphotericin B may be able to relieve fungal infection which can be a side effect of chemotherapy. Colony-stimulating factors such as sargramostim may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy. It is not yet known whether receiving liposomal amphotericin B plus sargramostim is more effective than receiving liposomal amphotericin B alone in treating patients with invasive fungal infection.

PURPOSE: Randomized double-blinded phase III trial to compare the effectiveness of liposomal amphotericin B with or without sargramostim in treating patients with invasive fungal infection.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the benefit of the cytokine sargramostim (GM-CSF) in resolving suspected or proven fungal infections in patients treated with systemic antifungal therapy (liposomal amphotericin B) who have been entered on protocols MRC-LEUK-AML11, AML12 or UKALLXII. II. Assess, in vitro, the effect of GM-CSF on monocyte function on cells taken from these patients.

OUTLINE: This is a double blind, supportive care study for patients on MRC-LEUK-AML11, AML12, or UKALLXII (or their successors). Patients are stratified according to proven or suspected fungal infection. Patients receive daily doses of intravenous liposomal amphotericin B based on stratification. All patients are then randomized to also receive either sargramostim (GM-CSF) (arm I) or a placebo (arm II) by subcutaneous injections (intravenous infusion over 4-6 hours is permitted if subcutaneous route is unacceptable). Treatment continues for 42 days. Some patients with localized lesions that clinically improve should be considered for surgical removal of the residual lesion. Patients may continue therapy after 42 days at the physician's discretion. Patients are assessed weekly until the end of study (particularly on day 28 and at end of study).

PROJECTED ACCRUAL: There will be 200 patients (100 in each arm) accrued into this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Patients entered into MRC-LEUK-AML11, AML12, UKALLXII, or their successors (including those undergoing bone marrow transplantation as part of the studies) who have a proven or suspected deep-seated fungal infection as listed below: Pulmonary fungal infection - proven or suspected Sinus infection - proven or suspected Fungemia - proven Chronic hepatosplenic candidosis - proven by CT/MRI Invasive cutaneous fungal infection - proven Cerebral fungal infection - proven or suspected

PATIENT CHARACTERISTICS: Age: 15 and over Performance status: Karnofsky 30-100% Life expectancy: At least 6 weeks Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No known intolerance to liposomal amphotericin B or sargramostim

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 3 months since sargramostim Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified Other: At least 2 weeks since liposomal amphotericin B

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 1997-07; Study Completion 1997-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C.H. Poynton, MD, Study Chair — University Hospital of Wales
Locations (1):
- University of Wales College of Medicine, Cardiff, Wales, United Kingdom